CLINICAL TRIAL: NCT00864695
Title: Role of Anesthesiologist-Patient Relationship in Changing Postoperative Perception of Patients Admitted to a Teaching Hospital
Brief Title: Role of Anesthesiologist-Patient Relationship
Status: Completed | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Faculdade de Medicina de Botucatu, UNESP, Botucatu, Brasil (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Clinical Research Ethics Committee of College of Medicine of Botucatu, College of Medicine of Botucatu
Other Study IDs: upeclin/HC/FMB-Unesp-21
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2009-03-19 (Estimated); Status verified 2009-03

CONDITIONS: Preoperative; Anesthesia; Postoperative
Keywords: Anesthesia; Ethics; Trends; Manpower; Perioperative care
MeSH Terms: interventions — Palliative Care; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Surgical patients: Individuals who were hospitalized in the Botucatu Medical School Hospital to undergo surgery under anesthesia administered by the Anesthesiology Service of BMS Department of Anesthesiology.
  Interventions: Other: Supportive care

INTERVENTIONS:
Other: Supportive care — protocol designed to evaluate one or more interventions where the primary intent is to maximize comfort, minimize side effects or mitigate against a decline in the subject's health or function. In general, supportive care interventions are not intended to cure a disease.
  Other Names: Questionnaire

SUMMARY:
Descriptive analytic survey of 1137 and 518 patients aged 16 years or more before and after anesthesia exposure, respectively to assess the anesthesiologist-patient relationship role on patient postoperative perception of the binominal anesthesia-anesthesiologist. The aim of this study was to assess the anesthesiologist-patient relationship role on patient postoperative perception of the binominal anesthesia-anesthesiologist.

Period: may/2007 to may/2008

DETAILED DESCRIPTION:
A questionnaire was used to determine patient characteristics and perception of anesthesia/anesthesiologist, as well as fears and concerns related to anesthesia. This descriptive-analytic study was based on opinions and information provided before and after anesthesia by individuals who were hospitalized in the Botucatu Medical School (BMS) Hospital to undergo surgery under anesthesia administered by the Anesthesiology Service of BMS Department of Anesthesiology. A questionnaire including structured questions aimed at determining patient characteristics (age, gender, race, marital status, education level, birthplace, provenance, surgical service of origin, occupation, history of anesthesia exposure) and perceptions of anesthesiologists/anesthesia, as well as open-ended questions that allowed respondents to add free comments, recorded as spoken, about their concerns before and after anesthesia. The post-anesthesia interview also included questions regarding the administration of pre-anesthetic drugs, recall of the anesthesiologist in the operating room, satisfaction with the care provided by the anesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

* conscious surgical patients
* 16 years or more
* Portuguese-speaking patients

Exclusion Criteria:

* patients with altered states of consciousness or expression/comprehension impairment
* patients who did not undergo anesthesia/surgery (cancelled or postponed)

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This descriptive-analytic study was based on opinions and information provided before and after anesthesia by individuals who were hospitalized in the Botucatu Medical School Hospital to undergo surgery under anesthesia. A questionnaire was used to determine patient characteristics and perception of anesthesia/anesthesiologist, as well as fears and concerns related to anesthesia.
Sampling Method: Probability Sample
Enrollment: 1137 (Actual)
Dates: Start 2007-05; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Role of anesthesiologist-patient relationship in changing postoperative perception of patients admitted to a teaching hospital | one year

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Leite, Principal Investigator — College Study of Medicine
Locations (1):
- College of Medicine of Botucatu, Botucatu, São Paulo, Brazil